CLINICAL TRIAL: NCT04956380
Title: Self-assessment Triage in Inflammatory Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Mary Bell, Rheumatologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 261-2017
Record Dates: First submitted 2018-04-11; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Arthritis
Keywords: New Referrals; Triage; Self-assessment
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Intervention Model Description: 2x2 factorial randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Joint Count + Early Inflammatory Arthritis Detection Tool (Experimental): Rheumatologist reviews both the self-administered tender joint count (out of 68 joints on a homunculus) and self-administered Early Inflammatory Arthritis Detection Tool that were completed by the patient. Rheumatologist then uses the information provided in these tools by the patient to determine whether they should advance the urgency rating of the case.
  Interventions: Other: Self-administered Triage
- Early Inflammatory Arthritis Detection Tool (Experimental): Rheumatologist reviews both the self-administered Early Inflammatory Arthritis Detection Tool that was completed by the patient. Rheumatologist then uses the information provided in this tool by the patient to determine whether they should advance the urgency rating of the case.
  Interventions: Other: Self-administered Triage
- Joint Count (Experimental): Rheumatologist reviews both the self-administered Patient Tender Joint Count that was completed by the patient. Rheumatologist then uses the information provided in this tool by the patient to determine whether they should advance the urgency rating of the case.
  Interventions: Other: Self-administered Triage
- Control (No Intervention): Rheumatologist does not review any of the self-administered tools completed by the patient.

INTERVENTIONS:
Other: Self-administered Triage — Self-assessment including a self-administered patient joint count and a self-administered Early Inflammatory Arthritis Detection Tool
  Arms: Early Inflammatory Arthritis Detection Tool; Joint Count; Joint Count + Early Inflammatory Arthritis Detection Tool

SUMMARY:
There are benefits to early, intensive treatment of IA. But getting to treatment depends on timeline and accurate case identification. The longest delays occur in persons self-identifying the need to see care for IA, recognition of these cases by primary care providers (PCPs), and appropriate, timely referral to rheumatology. Current methods of improving time to referral and consultation are effective, but costly and unsustainable, so there is need to look for alternatives. One solutions may be the use of patient self-administered tools.

In this study, we will test whether the use of validated, self-administered patient questionnaires (self-assessment) can advance the urgency rating of referrals for people with inflammatory arthritis (IA). If urgency ratings can be advanced then self-assessment may have the potential to reduce wait times to see a rheumatologist.

In Canada, one in every hundred people has IA and hundreds of new patients are diagnosed each year. Wait times to see a rheumatologist are long, so anything that has the potential to reduce these wait times would have a significant impact.

ELIGIBILITY:
Inclusion Criteria:

* new patient referral

Exclusion Criteria:

* under 18 years of age
* confirmed diagnosis of inflammatory condition
* seen/managed by another rheumatologist within the last five years
* unable to speak English
* on disease modifying antirheumatic drugs.
* referrals from the Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Urgency Rating | 1 Day
  When a rheumatologist receives a new referral, he/she gives it an "urgency rating", which indicates how soon the patient needs to be seen based on information they have about the patient in the referral letter. Urgency rating has four levels: 1) urgent, schedule patient within 4 weeks, 2) urgent, schedule patient in 4 to 6 weeks, 3) urgent, schedule patient in 6 to 12 weeks, 4) non-urgent, schedule patient after 12 weeks. These were developed by the Canadian Rheumatology Association. Please note that these are NOT time points, but ratings used to describe how soon a patient should be seen.
  Urgency rating will be recorded by the rheumatologist after three different cases: 1) After the rheumatologist receives the patient's referral letter, 2) after the patient arrives for their first appointment and completes a self-assessment in the waiting area, and 3) after the rheumatologist completes their first physical assessment of the patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dr. Raheem Kherani, Richmond, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be faxed from Richmond Site to Toronto Site for entry and analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data is currently being collected and faxed. Data will remain available for 10 years.